CLINICAL TRIAL: NCT07323303
Title: Real-World Study on the Burden of Hidradenitis Suppurativa
Status: Not yet recruiting | Type: Observational
Sponsor: PeriPharm (Other)
Responsible Party: Sponsor
Other Study IDs: PROxy85HS
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with HS: Patient diagnosed with HS
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No specific intervention is assess in this study. Observational cohort.

SUMMARY:
Despite the significant impact of HS on patients' quality of life (QoL) and daily functioning, there remains limited real-world evidence describing the burden of this condition in Canada. HS is an under-recognized and often misdiagnosed condition, with a substantial psychological and physical burden on patients. Understanding the real-world experiences of individuals living with HS in Canada can help identify unmet needs and inform patient-centered care approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with HS;
2. Aged ≥18 years;
3. Able to read and understand French or English;
4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Participation in an interventional study for HS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with HS
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To estimate work productivity loss in patients with HS. | At recruitment
  Using the Work Productivity and Activity Impairment (WPAI) questionnaire. This questionnaire provides a quantitative measure of impairment over the last 7 days and includes four metrics: absenteeism (work time missed because of health issues during the past 7 days), presenteeism (impairment while working due to health issues during the past 7 days), overall work productivity loss (combination of absenteeism and presenteeism), and activity impairment.

SECONDARY OUTCOMES:
To estimate the QoL of patients with HS | At recruitment
  The Hidradenitis Suppurativa Quality of Life Questionnaire (HiSQOL) is a validated, HS-specific instrument designed to capture the multidimensional impact of HS on quality of life over the previous 7 days. It consists of 17 items that use Likert-type response options, ranging from 0 ("not at all") to 4 ("extremely"), with some items allowing respondents to indicate that an activity was not performed due either to lack of relevance or HS severity
To estimate pain intensity in patients with HS. | At recruitment
  Patients with HS will self-report the worst intensity of their pain over the past 7 days using an 11-point numeric rating scale (NRS). The NRS ranges from 0 ("No Pain") to 10 ("The worst imaginable Pain"). Pain was selected as a key symptom given its substantial impact on patients' daily lives and QoL. The 7-day recall period was chosen to balance recall accuracy and symptom variability, capturing recent disease activity while minimizing recall bias.

IPD SHARING:
Plan to Share IPD: No